CLINICAL TRIAL: NCT03352232
Title: Oxygenating the Potential: Hyperbaric Oxygen and Manipulative Therapies to Regain Function in Stroke Survivors
Brief Title: Hyperbaric Oxygen and Manipulative Therapies to Regain Function Post Stroke
Acronym: HBOT/OMT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abington Memorial Hospital (Other)
Collaborators: Philadelphia College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Hana Choe, Assistant Director NeuroIntervention and Neurocritical Care, Abington Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-063
Record Dates: First submitted 2017-11-14; First posted 2017-11-24 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Stroke; Motor Dysfunction; Chronic Stroke; Ischemic Stroke
MeSH Terms: conditions — Stroke; Neurologic Manifestations; Ischemic Stroke | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: There will be two populations based on when they experienced a stroke. Subacute stroke patients will have suffered an ischemic stroke within 3 months of enrollment and have persistent neurological deficits. The second group will be patients who suffered an ischemic stroke more than 6 months (chronic) from time of enrollment and have persistent neurological deficits compromising activities of daily living.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subacute Ischemic Stroke (Experimental): Subacute stroke patients post stroke within 3 months of enrollment, have persistent neurological deficits despite conventional rehabilitation
  Interventions: Combination Product: HBOT and OMT
- Chronic Ischemic Stroke (Experimental): Chronic stroke patients more than 6 months from stroke with persistent neurological deficits despite conventional rehabilitation
  Interventions: Combination Product: HBOT and OMT

INTERVENTIONS:
Combination Product: HBOT and OMT — Hyperbaric oxygen therapy (HBOT) is defined as breathing 100% oxygen at increased atmospheric pressure. Osteopathic manipulative therapy (OMT) is used for myriad ailments including contractures, pain, spasticity. Patients in intervention arms will receive hyperbaric oxygen therapy at 2ATM (atmospheres) for 90minutes daily for up to 6weeks. In addition, they will receive osteopathic manipulative therapies twice a week during the same treatment phase.
  Other Names: Osteopathic manipulative therapies (OMT); Hyperbaric Oxygen Therapy (HBOT)

SUMMARY:
To study safety, feasibility and outcomes of combining osteopathic manipulative therapies with hyperbaric oxygen therapy in reducing the functional deficits in stroke survivors in subacute and chronic phases post ischemic stroke. To document the same as part of a pilot project in anticipation of further investigational studies.

DETAILED DESCRIPTION:
The primary objective of this study is to show that hyperbaric oxygen therapy combined with osteopathic manipulative therapies improve outcomes in patients who have persistent neurological deficits after ischemic stroke compared to historical norms.

The secondary objectives of this study is to demonstrate safety and feasibility of treating patients post stroke with hyperbaric oxygen and osteopathic therapies as well as determine improvements in multiple assessment scales of motor function, depression, activities of daily living(ADL) and pain

ELIGIBILITY:
Inclusion Criteria:

1. Post Ischemic stroke
2. Patients aged 18-80
3. NIHSS >5
4. mRS>/=3, which connotes moderate disability requiring some help.
5. Persistent significant motor dysfunction of at least one arm
6. Subacute stroke patients (within three months from time of stroke)
7. Chronic stroke patients (more than 6months from time of stroke)
8. Patient must be able to understand instructions and verbalize discomfort
9. Reliable attendance for daily (M-F) HBOT treatment and 2x/week OMT sessions for up to 6weeks

Exclusion Criteria:

1. Hemorrhagic stroke
2. Prior functional disability mRS >1
3. Expressive or receptive aphasia
4. Bedbound patients due to lifting limitations for HBOT
5. History of severe, advanced emphysema with bullous disease
6. Prior history of spontaneous pneumothorax or chest surgery
7. Prior history of depression requiring medications
8. Pregnancy
9. Concomitant non-conventional rehab therapies including: acupuncture, botulinum toxin injections, massage therapy
10. Significant claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
National Institute of Health Stroke Score (NIHSS) 0-5 or Modified Rankin Score (mRS) 0-2 | 90 Days
  Primary Outcome NIHSS 0-5, 0 without deficits; mRS 0-2, 0 without disability - 2 slight disability, no need for assistance

SECONDARY OUTCOMES:
Beck Depression Inventory | 90 days
  assessment of Depression scale rating
Wolf Motor Score | 90 days
  assessment of functional motor recovery
Rivermead Extended Activities of Daily Living (EADL) scale | 90 days
  assessment of capability navigating usual and community based ADLs
Medical Outcomes 36 Item | 90 days
  assessment of global health
Functional Independence Measure (FIM) | 90 days
  universally used assessment of patient's ability to perform activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Hana Choe, MD, Principal Investigator — Abington Memorial Hospital
Locations (1):
- Abington Memorial Hospital, Abington, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No